CLINICAL TRIAL: NCT03381781
Title: Decitabine,Cytarabine(Ara-C) and Arsenic Trioxide(ATO) in the Treatment of Acute Myeloid Leukemia With p53 Mutations
Brief Title: Decitabine,Cytarabine and Arsenic Trioxide for Acute Myeloid Leukemia With p53 Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Li Junmin (Other)
Responsible Party: Sponsor-Investigator, Li Junmin, director of the hematology department, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RuijinH mutant p53 AML
Record Dates: First submitted 2017-11-21; First posted 2017-12-22 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Acute Myeloid Leukemia; P53 Mutation
Keywords: p53 mutation; acute myeloid leukemia; decitabine; Arsenic trioxide; cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Arsenic Trioxide; Arsenic; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients with p53 mutations will be treated with Decitabine,Arsenic Trioxide and Cytarabine.
  Interventions: Drug: Decitabine; Drug: Arsenic Trioxide; Drug: Cytarabine

INTERVENTIONS:
Drug: Decitabine — 20mg/m^2,d1-5,ivgtt,28days as a duration
  Other Names: DNA demethylation agent; DNA damaging agent
Drug: Arsenic Trioxide — 0.16mg/kg,d1-5,ivgtt,28days as a duration
  Other Names: As2O3; Arsenic
Drug: Cytarabine — 15mg/m^2,hypodermic injection,q12h,d1-7
  Other Names: DNA damaging agent; Ara-C

SUMMARY:
This is a prospective,uncontrolled and multi-institution trial.The aim is to identify if using decitabine,cytarabine and ATO as the therapy of acute myeloid leukemia(AML) with p53 mutations has better relapse free survival and complete response than using decitabine and cytarabine.

TP53 mutation is commonly associated with poor cancer patient prognosis yet no mutant p53 (mp53)-targeting regimen was clinically established. Particularly, p53 mutation is associated with extremely poor prognosis in myelodysplastic syndromes (MDS) and acute myeloid leukemia (AML) patients.

Decitabine (DAC) is a FDA approved drug for MDS treatment. In two independent clinical trials reported recently, DNA demethylating drug DAC treatment yielded a surprisingly high rate of complete remission (CR) in mp53-harboring AML/MDS patients (Welch, NEJM, 2016; Chang, BJH, 2017). Notably, all of the mp53-expressing patients in the two clinical studies relapsed quickly.

Arsenic trioxide (ATO) is a FDA approved drug for M3-AML treatment. Despite of the observed efficacy in treating non-APL patients, ATO is not yet approved for non-APL cancer treatment. ATO plays key role in regulating both wild-type p53 (wtp53) and mp53. Our published and unpublished data suggest ATO potentially hijacks nuclear iASPP-mediated STRaND pathway via exposing iASPP's RaDAR nuclear import code (Lu, Cancer Cell, 2013; Lu, Cell, 2014; Lu, Nat Rev Mol Cell Biol, 2016; Lu, unpublished). Our unpublished data also suggests a key role of ATO in regulating mp53 (Lu, The 17th International p53 Workshop, 2017). ATO is widely reported to be able to degrade and thus inhibit mp53's oncogenic function (Hamadeh, BBRC, 1999)(Liu, Blood, 2003). ATO suppressed cancer cell growth by targeting mp53 for degradation by Pirh2 degradation pathway (Yang, JBC, 2011; Yan, PLOS one, 2014);

Here we explore the potential of combination of DAC and ATO in improving the mp53-harboring AML/MDS patients' relapse free survival (RFS) and the ability to thoroughly eliminate mp53 subclone. Basic researches aiming to explore the mechanisms how mp53 cells responds to DAC and/or ATO treatment and how mp53 cells develop resistance to DAC and/or ATO will be coupled. We designate trials aiming for a better treatment regimen for mp53 patients as 'PANDA-Trials'.

DETAILED DESCRIPTION:
This study is designed as a model of precision medicine. About 1500 AML patients will be applied for TP53 sequencing. The bone marrow samples will be collected and its p53 status will be Sanger sequenced in 3-5 days before drug administration. The 100 mp53-positive patients will be trialed, while the others (mp53-negative patients) will be subjected to standard treatment or other clinical trials.

In this study,100 patients with p53 mutations will be enrolled,including newly diagnosed AML aged 60-75,AML transferred from Myelodysplastic Syndrome(MDS) and therapy related AML.

ELIGIBILITY:
Inclusion Criteria:

* de novo elderly AML,AML transferred from MDS,therapy related AML
* exclude acute promyelocytic leukemia(APL)
* p53 mutations determined by DNA sequencing from bone marrow
* ECOG<3,CCI≤1,ADL≥100
* bone marrow is active
* normal hepatic function and renal function
* normal cardiac function
* obtain informed consent

Exclusion Criteria:

* APL
* without p53 mutations
* previously treated elderly AML
* central nervous system is involved
* abnormal hepatic function or renal function
* severe cardiac disease,including myocardial infarction,cardiac dysfunction
* ECG:QTc>0.44 sec in men,QTc>0.46 sec in women
* with other malignant tumor meanwhile
* active tuberculosis or HIV-positive patients
* woman who are pregnant or breastfeeding
* allergic to any drug in protocol or with contraindications
* hypomethylation agent(HMA) is contraindicated
* ECOG≥3,CCI>1,ADL<100
* cannot understand or obey the protocol
* with a history of allergies or intolerability
* with a history of decitabine therapy
* participate in other clinical trials meanwhile
* any situations that hinder trial existed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
relapse free survival | From date of complete release until the date of first documented relapse, assessed up to 6-8months
  since a patient first being determined as complete release until relapse

SECONDARY OUTCOMES:
complete release | 2-4 months since the first cycle of treatment
  the percent of patients with complete release in all patients enrolled
overall survival | primary estimated for 1year
  from first diagnosed to death whichever the cause is

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Sujiang, Principal Investigator — Shanghai Ruijin Hospital North; Lu Min, Principal Investigator — Shanghai institute of Hematology
Locations (3):
- China (3):
  - Ruijin Hospital North, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai Institute of Hematology, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang CK, Zhao YS, Xu F, Guo J, Zhang Z, He Q, Wu D, Wu LY, Su JY, Song LX, Xiao C, Li X. TP53 mutations predict decitabine-induced complete responses in patients with myelodysplastic syndromes. Br J Haematol. 2017 Feb;176(4):600-608. doi: 10.1111/bjh.14455. Epub 2016 Dec 16. PMID 27984642
- [Background] Welch JS, Petti AA, Miller CA, Fronick CC, O'Laughlin M, Fulton RS, Wilson RK, Baty JD, Duncavage EJ, Tandon B, Lee YS, Wartman LD, Uy GL, Ghobadi A, Tomasson MH, Pusic I, Romee R, Fehniger TA, Stockerl-Goldstein KE, Vij R, Oh ST, Abboud CN, Cashen AF, Schroeder MA, Jacoby MA, Heath SE, Luber K, Janke MR, Hantel A, Khan N, Sukhanova MJ, Knoebel RW, Stock W, Graubert TA, Walter MJ, Westervelt P, Link DC, DiPersio JF, Ley TJ. TP53 and Decitabine in Acute Myeloid Leukemia and Myelodysplastic Syndromes. N Engl J Med. 2016 Nov 24;375(21):2023-2036. doi: 10.1056/NEJMoa1605949. PMID 27959731
- [Background] Lu M, Breyssens H, Salter V, Zhong S, Hu Y, Baer C, Ratnayaka I, Sullivan A, Brown NR, Endicott J, Knapp S, Kessler BM, Middleton MR, Siebold C, Jones EY, Sviderskaya EV, Cebon J, John T, Caballero OL, Goding CR, Lu X. Restoring p53 function in human melanoma cells by inhibiting MDM2 and cyclin B1/CDK1-phosphorylated nuclear iASPP. Cancer Cell. 2013 May 13;23(5):618-33. doi: 10.1016/j.ccr.2013.03.013. Epub 2013 Apr 25. PMID 23623661
- [Background] Lu M, Muers MR, Lu X. Introducing STRaNDs: shuttling transcriptional regulators that are non-DNA binding. Nat Rev Mol Cell Biol. 2016 Aug;17(8):523-32. doi: 10.1038/nrm.2016.41. Epub 2016 May 25. PMID 27220640
- [Background] Lu M, Zak J, Chen S, Sanchez-Pulido L, Severson DT, Endicott J, Ponting CP, Schofield CJ, Lu X. A code for RanGDP binding in ankyrin repeats defines a nuclear import pathway. Cell. 2014 May 22;157(5):1130-45. doi: 10.1016/j.cell.2014.05.006. PMID 24855949
- [Background] Yan W, Jung YS, Zhang Y, Chen X. Arsenic trioxide reactivates proteasome-dependent degradation of mutant p53 protein in cancer cells in part via enhanced expression of Pirh2 E3 ligase. PLoS One. 2014 Aug 12;9(8):e103497. doi: 10.1371/journal.pone.0103497. eCollection 2014. PMID 25116336